CLINICAL TRIAL: NCT02484794
Title: Efficacy and Acceptability of Augmenting Specialty Eating Disorder Clinical Treatment With a Smartphone Application: A Pilot RCT
Brief Title: Augmenting Specialty Eating Disorder Clinical Treatment With a Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59093007
Record Dates: First submitted 2015-06-23; First posted 2015-06-30 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Eating Disorders
Keywords: Eating Disorders; Smartphone; App; Mobile Health; Recovery Record; Cognitive Behavioural Therapy; Outpatient Program; Self Monitoring
MeSH Terms: conditions — Feeding and Eating Disorders; Alzheimer Disease | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (Active Comparator): Patients will receive standard outpatient treatment that consists of group psychotherapy, skills training, self-monitoring, nutritional counselling, and meal support.
  Interventions: Behavioral: Standard Outpatient Treatment
- Treatment with Smartphone App (Experimental): Patients will receive the same standard outpatient treatment but will use the smartphone application instead of the paper food record. Patients in this group will receive daily feedback through the app, as opposed to weekly, but will still attend the weekly nutritional counselling group.
  Interventions: Behavioral: Standard Outpatient Treatment; Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Standard Outpatient Treatment — Standard treatment offered by the Nova Scotia Health Authority Eating Disorder Outpatient Program varies in intensity but involves therapy groups (e.g., goal setting and skill building groups), individual contact, and meal experiences. Minimal participation in the program consists of a weekly nutritional counselling group (Nutri-Logical) and one supervised meal a week. In the nutritional counselling group, patients keep a food journal (self-monitor), set eating goals, receive feedback from a psychologist and dietitian, and share experiences with the group.
  Other Names: Treatment as Usual (TAU)
Behavioral: Smartphone App — The smartphone app is a mobile eating disorder self-monitoring tool that incorporates discrete reminders, positive feedback, social support, summative feedback, coping skill suggestions, and linking patients with their treating clinicians (psychologist and dietician). The app is CBT-based and was designed as an alternative to paper food records for use in clinical treatment.
  Other Names: Recovery Record App
  Arms: Treatment with Smartphone App

SUMMARY:
Cognitive behavioural therapy (CBT) is the most empirically supported and researched treatment for eating disorders. A central component of CBT for eating disorders is self-monitoring which involves patients keeping a paper food record of their meals and associated thoughts, feelings, and behaviours and receiving feedback from a clinician to help target dysfunctional cognitions and behaviours. Given the issues associated with paper journals such as non-compliance, feelings of shame when used in public, and delayed feedback, researchers have developed an evidence-based smartphone application (Recovery Record) for eating disorder self-monitoring that links patients with their clinicians and offers additional features designed to enhance treatment.

The current pilot randomised controlled trial (RCT) seeks to evaluate this smartphone application in a clinical setting alongside standard eating disorder outpatient treatment. Patients will be recruited from the Nova Scotia Health Authority Eating Disorder Outpatient Program and randomised to receive either standard treatment or standard treatment with the app (instead of the paper food record). The efficacy and acceptability of both treatments will be assessed and compared. Coping skill use and self-efficacy among patients will also be examined given the skill building focus of treatment and in-app capabilities to deliver real-time coping skill suggestions to patients.

This pilot study will be the first to examine the efficacy and acceptability of a smartphone application in eating disorder clinical treatment and if successful, should provide preliminary support for the use of smartphone applications over traditional paper food journals as a self-monitoring tool for augmenting specialty eating disorder clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an eating disorder (anorexia nervosa, bulimia nervosa, or eating disorder not otherwise specified) according to DSM-V criteria (American Psychiatric Association, 2013) as determined through a standard clinical interview by either a team psychiatrist or clinical psychologist, and validated with a self-report diagnostic measure.
* Patients with an Apple or Android smartphone (a mobile phone with access to third-party applications and advanced features) with an active data plan or frequent (e.g., daily) Wi-Fi access.
* Patients 17 years or older.
* Signed consent from patient.

Exclusion Criteria:

* Patient has insufficient knowledge of English.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in eating disorder severity as assessed by the Eating Disorder Examination Questionnaire (EDE-Q) | Pre-treatment, 2 months, post-treatment (up to 8 months after pre-treatment), 3-month follow-up
  A self-report scale that assesses the severity of 4 areas of eating disorder pathology: Eating Concern, Weight Concern, Dietary Restraint, and Shape Concern. Overall eating disorder severity is also assessed.

SECONDARY OUTCOMES:
Change in coping skill use as assessed by the Cognitive Behavioral Therapy Skills Questionnaire (CBTSQ) | Pre-treatment, 2 months, post-treatment (up to 8 months after pre-treatment), 3-month follow-up
  A self-report measure that assesses the use of CBT-taught skills.
Change in coping skill use as assessed by the Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) | Pre-treatment, 2 months, post-treatment (up to 8 months after pre-treatment), 3-month follow-up
  A self-report measure that assesses the use of DBT-taught coping skills and dysfunctional coping skills.
Change in coping self-efficacy as assessed by the Coping Self-Efficacy Scale (CSES) | Pre-treatment, 2 months, post-treatment (up to 8 months after pre-treatment), 3-month follow-up
  A self-report scale that assesses confidence in using various coping skills.
Treatment acceptability as assessed by the Outpatient Client Experience Survey | Post-treatment (up to 8 months after pre-treatment)
  A questionnaire of overall experiences with a mental health or addictions tertiary outpatient program.
Treatment acceptability as assessed by a treatment-specific questionnaire | Post-treatment (up to 8 months after pre-treatment)
  Additional Likert scale/open-ended questions pertaining to the self-monitoring tool used (app or paper food record) were developed to assess patient satisfaction with treatment (e.g., "I felt that I could discretely log my meals.").
Dropout rate | Post-treatment (up to 8 months after pre-treatment)
  Dropout rates will be calculated for each group as a measure of treatment acceptability.

OTHER OUTCOMES:
Diagnoses validated by the Eating Disorder Diagnostic Scale (EDDS) | Pre-treatment
  A self-report diagnostic measure that will be used to validate clinical diagnoses (as determined by team psychiatrist or clinical psychologist).

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Keshen, MD, FRCPC, Principal Investigator — Nova Scotia Health Authority/Dalhousie University
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Keshen A, Helson T, Ali S, Dixon L, Tregarthen J, Town J. Efficacy and acceptability of self-monitoring via a smartphone application versus traditional paper records in an intensive outpatient eating disorder treatment setting. Eur Eat Disord Rev. 2020 Jul;28(4):473-479. doi: 10.1002/erv.2727. Epub 2020 Feb 12. PMID 32050044